CLINICAL TRIAL: NCT00392730
Title: Neurodevelopment and Neuroimaging in Parenterally-fed Infants and Young Children
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Principal Investigator, Judy Aschner, Adjunct Professor of Pediatrics, Vanderbilt University
Other Study IDs: Gerber07-01-06JLA; ES013730
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Parenteral Nutrition; Necrotizing Enterocolitis; Digestive System Abnormalities; Cholestasis
Keywords: Manganese; Neonatal Intensive Care; MRI; Parenteral Nutrition; Prematurity
MeSH Terms: conditions — Hyperphagia; Enterocolitis, Necrotizing; Digestive System Abnormalities; Cholestasis; Premature Birth

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Preterm infants in NICU and age-matched controls
  Interventions: Dietary Supplement: Remove Mn from PN if evidence of increased brain Mn on MRI
- 2: Term infants in NICU and age-matched controls
  Interventions: Dietary Supplement: Remove Mn from PN if evidence of increased brain Mn on MRI
- 3: Children on home PN (to age 6) and age-matched controls
  Interventions: Dietary Supplement: Remove Mn from PN if evidence of increased brain Mn on MRI

INTERVENTIONS:
Dietary Supplement: Remove Mn from PN if evidence of increased brain Mn on MRI — Withhold Mn-containing trace element cocktail and add zinc, copper and chromium individually to PN

SUMMARY:
Manganese (Mn) is an essential metal required for normal growth and development. However, exposure to high Mn levels can be toxic to the brain. The objectives of this project are to identify neonatal and young pediatric populations that are at increased risk of excessive brain Mn deposition and altered cognitive and motor development based on their dietary parenteral Mn exposure, and to make sound and evidence-based recommendations for appropriate Mn supplementation and monitoring of infants and young children receiving parenteral nutrition (PN). Our studies are designed to test the hypotheses that, compared with unexposed age-matched controls, infants and young children receiving prolonged Mn-supplemented PN will have increased deposition of Mn in their brains and lower scores on neurodevelopmental, cognitive and psychophysiological assessments.

DETAILED DESCRIPTION:
Specific Aims have been designed to test these hypotheses in three developmentally distinct populations:

1. preterm infants and
2. full term infants in the Neonatal Intensive Care Unit (NICU) requiring prolonged PN and
3. older infants and young children on home PN.

Mn neurotoxicity will be investigated by longitudinal assessments of cognitive (executive functioning battery), neurodevelopmental (Bayley III Scales of Infant Development), and psychophysiological (event-related potential) measures and will be correlated with brain deposition of Mn using the technique of magnetic resonance (MR) relaxometry in a vulnerable population of infants receiving Mn-supplemented PN and age-matched controls. This proposal addresses a clinically relevant and unexplored link between nutritional practices, brain Mn deposition and neurodevelopmental sequelae in an at-risk population of infants and young children utilizing state-of-the-art magnetic resonance imaging (MRI) technology and neurodevelopmental assessment techniques. The potential for increased brain Mn accumulation in infants, and by inference, the potential health risks associated with elevated brain Mn burden, represents crucial, unexplored issues of exposure and susceptibility. The potential contribution of Mn toxicity to the poor outcomes of infants dependent for an extended time on PN has not been fully acknowledged or studied. Improved understanding of the relationships between Mn exposure and developmental outcomes will undoubtedly lead to altered clinical practices and more careful monitoring of Mn intake and blood and/or brain Mn levels in high risk infants. Our studies will also contribute to an improved understanding of the value of non-invasive MR imaging in the monitoring of pediatric patients on PN.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than 30 days postnatal age
2. In the preceding four weeks, have received >75% of their nutrition as Mn-supplemented PN
3. Clinically stable for transport to the MR facility
4. Signed parental consent.

Or healthy age-matched controls

Exclusion Criteria:

1. Any infant not expected to survive to the age of 3 months or
2. Not expected to achieve sufficient clinical stability to tolerate the MRI procedure.

Ages: 30 Days to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Term and preterm infants on prolonged PN in the NICU and post-discharge and young children on home PN and age-matched controls
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2006-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Brain Mn deposition measured by MR relaxometry | baseline (at study enrolment)
  Mn neurotoxicity will be investigated by magnetic resonance (MR) relaxometry in a population of infants receiving Mn-supplemented parenteral nutrition and age-matched controls.

SECONDARY OUTCOMES:
Neurodevelopmental outcomes | 2 years
  Neurodevelopment will be investigated by longitudinal assessments of cognitive (executive functioning battery), neurodevelopmental (Bayley III Scales of Infant Development), and psychophysiological (event-related potential) measures

CONTACTS AND LOCATIONS:
Overall Officials: Judy L Aschner, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Children's Hospital, Nashville, Tennessee, United States

REFERENCES:
- [Background] Aschner JL, Aschner M. Nutritional aspects of manganese homeostasis. Mol Aspects Med. 2005 Aug-Oct;26(4-5):353-62. doi: 10.1016/j.mam.2005.07.003. PMID 16099026
- [Background] Fitsanakis VA, Zhang N, Avison MJ, Gore JC, Aschner JL, Aschner M. The use of magnetic resonance imaging (MRI) in the study of manganese neurotoxicity. Neurotoxicology. 2006 Sep;27(5):798-806. doi: 10.1016/j.neuro.2006.03.001. Epub 2006 Apr 18. PMID 16620989
- [Background] Fitsanakis VA, Piccola G, Marreilha dos Santos AP, Aschner JL, Aschner M. Putative proteins involved in manganese transport across the blood-brain barrier. Hum Exp Toxicol. 2007 Apr;26(4):295-302. doi: 10.1177/0960327107070496. PMID 17615110
- [Background] Yin Z, Aschner JL, dos Santos AP, Aschner M. Mitochondrial-dependent manganese neurotoxicity in rat primary astrocyte cultures. Brain Res. 2008 Apr 8;1203:1-11. doi: 10.1016/j.brainres.2008.01.079. Epub 2008 Feb 11. PMID 18313649
- [Derived] Aschner JL, Anderson A, Slaughter JC, Aschner M, Steele S, Beller A, Mouvery A, Furlong HM, Maitre NL. Neuroimaging identifies increased manganese deposition in infants receiving parenteral nutrition. Am J Clin Nutr. 2015 Dec;102(6):1482-9. doi: 10.3945/ajcn.115.116285. Epub 2015 Nov 11. PMID 26561627